CLINICAL TRIAL: NCT02858180
Title: A Multicenter, Open-label Study of Harvoni ® (Sofosbuvir Ledipasvir Fixed Dose Combination) in Subjects Infected With Chronic Hepatitis C and Advanced Heart Failure or Lung Disease
Brief Title: Hepatitis C Virus(HCV) Heart and Lung Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00069602
Record Dates: First submitted 2016-08-01; First posted 2016-08-08 (Estimated); Results first posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis C, Chronic; Heart Failure; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial
MeSH Terms: conditions — Hepatitis C, Chronic; Heart Failure; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial | interventions — Sofosbuvir; ledipasvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heart Failure Cohort (Experimental): Harvoni (sofosbuvir/ledipasvir fixed dose combination)
  1 pill once daily Includes 400 mg sofosbuvir (SOF) and 90 mg ledipasvir (LDV)
  Interventions: Drug: Sofosbuvir/ledipasvir fixed dose combination(SOF/LDV FDC)
- Lung Disease Cohort (Experimental): Harvoni (sofosbuvir/ledipasvir fixed dose combination)
  1 pill once daily Includes 400 mg sofosbuvir and 90 mg ledipasvir
  Interventions: Drug: Sofosbuvir/ledipasvir fixed dose combination(SOF/LDV FDC)

INTERVENTIONS:
Drug: Sofosbuvir/ledipasvir fixed dose combination(SOF/LDV FDC) — 1 pill once daily of SOF/LDV FDC
  Other Names: Harvoni

SUMMARY:
This is a multicenter study in Hepatitis C Virus (HCV) infected adult patients who also have advanced cardiac disease or advanced lung disease.

DETAILED DESCRIPTION:
This is a multicenter study in HCV infected adult patients who also have either advanced cardiac disease, or advanced lung disease. Advanced cardiac disease is defined as a marked limitation of physical activity, or discomfort upon physical activity. The patients in the advanced cardiac disease group must also have been hospitalized for heart failure within the last 12 months.

Advanced lung disease is defined as patients who have been diagnosed with chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD). Patients in the COPD group must have abnormalities in their forced expiratory volume (FEV) test, which measures the amount of air exhaled. They may or may not need supplemental oxygen. Patients in the ILD group must have been diagnosed with ILD and require supplement oxygen at all times.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV Infection of Genotype 1, 4, 5, or 6
* HCV RNA > 103 IU/mL at screening
* 18 years of age or older
* Diagnosis of chronic HCV infection, defined as positive HCV antibody or HCV RNA more than 6 months prior to screening OR an assessment of fibrosis F2 or greater prior to screening.

Subjects in the advanced heart failure cohort must meet all HCV criteria, and all of the following criteria:

* New York Heart Association (NYHA) Class III or IV functional classification

  * NYHA Class III: Subjects with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation, dyspnea, or anginal pain.
  * NYHA Class IV: Patient with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
* ejection fraction ≤ 30%
* hospitalized for heart failure in last 12 months

Subjects in the advanced lung disease cohort must have been diagnosed with chronic obstructive pulmonary disease (COPD) or interstitial lung disease (ILD) must meet all HCV criteria, and meet the following criteria for COPD or ILD:

* ILD criteria: diagnosis of interstitial lung disease with chronic supplemental oxygen requirement at rest and/or with exertion.
* COPD criteria (one of the following):

  * Forced expiratory volume (FEV1)< 30% predicted
  * OR any FEV1 with chronic supplemental oxygen requirement at rest and/or with exertion
  * OR any FEV1 with chronic hypercapnia (baseline partial pressure of arterial carbon dioxide [PaCO2] > 45)

Exclusion Criteria:

* Chronic HCV Infection with Genotype 2 or 3
* Treatment with any of the following agents

  * Amiodarone. Subjects previously treated with amiodarone must have stopped the amiodarone at least 60 days prior to day 1 of SOF/LDV FDC
  * Carbamazepine, phenytoin, phenobarbital, oxcarbazepine
  * Rifabutin, rifampin or rifapentine
  * HIV regimens containing tenofovir or tipranavir/ritonavir
  * St. John's wort
  * Rosuvastatin
* Have any serious or active medical or psychiatric illness which, in the opinion of the investigator, would interfere with subject treatment, assessment, or compliance
* History of hepatic encephalopathy or variceal hemorrhage
* Hepatitis B surface antigen positive
* Abnormal hematological and biochemical parameters, including:

  * Hemoglobin (Hb) < 8 g/dL
  * Platelets ≤ 50,000/mm3
  * alanine aminotransferase (ALT), aspartase aminotransferase (AST), or alkaline phosphatase ≥ 10 times upper limit of normal(ULN)
  * Total bilirubin > 3 mg/dl
  * Severe renal impairment creatinine clearance (CrCl), i.e. < 30 mL/min.
* History of major organ transplantation with an existing functional graft.
* History of clinically-significant drug allergy to nucleoside/nucleotide analogs.
* Pregnant women or women planning to become pregnant
* Women who are breastfeeding
* Active or recent history (≤ 1 year) of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12; Primary Completion 2019-04-11 (Actual); Study Completion 2019-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Muir, MD, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center - Dept of Gastroenterology, Durham, North Carolina
  - Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Via manuscript

REFERENCES:
- [Background] Mohd Hanafiah K, Groeger J, Flaxman AD, Wiersma ST. Global epidemiology of hepatitis C virus infection: new estimates of age-specific antibody to HCV seroprevalence. Hepatology. 2013 Apr;57(4):1333-42. doi: 10.1002/hep.26141. Epub 2013 Feb 4. PMID 23172780
- [Background] Armstrong GL, Wasley A, Simard EP, McQuillan GM, Kuhnert WL, Alter MJ. The prevalence of hepatitis C virus infection in the United States, 1999 through 2002. Ann Intern Med. 2006 May 16;144(10):705-14. doi: 10.7326/0003-4819-144-10-200605160-00004. PMID 16702586
- [Background] Ghany MG, Strader DB, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C: an update. Hepatology. 2009 Apr;49(4):1335-74. doi: 10.1002/hep.22759. No abstract available. PMID 19330875
- [Background] Afdhal N, Zeuzem S, Kwo P, Chojkier M, Gitlin N, Puoti M, Romero-Gomez M, Zarski JP, Agarwal K, Buggisch P, Foster GR, Brau N, Buti M, Jacobson IM, Subramanian GM, Ding X, Mo H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Mangia A, Marcellin P; ION-1 Investigators. Ledipasvir and sofosbuvir for untreated HCV genotype 1 infection. N Engl J Med. 2014 May 15;370(20):1889-98. doi: 10.1056/NEJMoa1402454. Epub 2014 Apr 11. PMID 24725239
- [Background] Feld JJ, Kowdley KV, Coakley E, Sigal S, Nelson DR, Crawford D, Weiland O, Aguilar H, Xiong J, Pilot-Matias T, DaSilva-Tillmann B, Larsen L, Podsadecki T, Bernstein B. Treatment of HCV with ABT-450/r-ombitasvir and dasabuvir with ribavirin. N Engl J Med. 2014 Apr 24;370(17):1594-603. doi: 10.1056/NEJMoa1315722. Epub 2014 Apr 10. PMID 24720703
- [Background] Lee I, Localio R, Brensinger CM, Blumberg EA, Lautenbach E, Gasink L, Amorosa VK, Lo Re V 3rd. Decreased post-transplant survival among heart transplant recipients with pre-transplant hepatitis C virus positivity. J Heart Lung Transplant. 2011 Nov;30(11):1266-74. doi: 10.1016/j.healun.2011.06.003. Epub 2011 Jul 20. PMID 21764330
- [Background] Fagiuoli S, Minniti F, Pevere S, Farinati F, Burra P, Livi U, Naccarato R, Chiaramonte M. HBV and HCV infections in heart transplant recipients. J Heart Lung Transplant. 2001 Jul;20(7):718-24. doi: 10.1016/s1053-2498(01)00255-8. PMID 11448796
- [Background] Sahi H, Zein NN, Mehta AC, Blazey HC, Meyer KH, Budev M. Outcomes after lung transplantation in patients with chronic hepatitis C virus infection. J Heart Lung Transplant. 2007 May;26(5):466-71. doi: 10.1016/j.healun.2007.01.037. Epub 2007 Mar 26. PMID 17449415
- [Background] Afdhal N, Reddy KR, Nelson DR, Lawitz E, Gordon SC, Schiff E, Nahass R, Ghalib R, Gitlin N, Herring R, Lalezari J, Younes ZH, Pockros PJ, Di Bisceglie AM, Arora S, Subramanian GM, Zhu Y, Dvory-Sobol H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Sulkowski M, Kwo P; ION-2 Investigators. Ledipasvir and sofosbuvir for previously treated HCV genotype 1 infection. N Engl J Med. 2014 Apr 17;370(16):1483-93. doi: 10.1056/NEJMoa1316366. Epub 2014 Apr 11. PMID 24725238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 12/2016 and 12/2018, 15 subjects with chronic HCV and advanced heart failure or chronic HCV and lung disease were enrolled across 4 sites (academic medical centers in the US). Subjects all have genotype 1, 4, 5 or 6 HCV.
Groups:
- Heart Failure Cohort: Harvoni (sofosbuvir/ledipasvir fixed dose combination)
  1 pill once daily Includes 400 mg sofosbuvir (SOF) and 90 mg ledipasvir (LDV)
  Sofosbuvir/ledipasvir fixed dose combination(SOF/LDV FDC): 1 pill once daily of SOF/LDV FDC
- Lung Disease Cohort: Harvoni (sofosbuvir/ledipasvir fixed dose combination)
  1 pill once daily Includes 400 mg sofosbuvir and 90 mg ledipasvir
  Sofosbuvir/ledipasvir fixed dose combination(SOF/LDV FDC): 1 pill once daily of SOF/LDV FDC
Period: Overall Study
Arm/Group | Heart Failure Cohort | Lung Disease Cohort
Started | 10 | 5
Completed | 10 (Completed a 12-week course of therapy.) | 3 (Completed a 12-week course of therapy.)
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heart Failure Cohort | Lung Disease Cohort | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (7.5) | 59.4 (5.1) | 60.1 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Completed 24 Weeks of Therapy
Description: The primary safety endpoint is the number of subjects who complete a full course of therapy.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure Cohort | Lung Disease Cohort
Number analyzed (Participants) | 10 | 5
Participants | 0 | 1

2. Secondary Outcome: Number of Subjects With Sustained Virologic Response (SVR) 12
Description: The secondary outcome of efficacy will be determined by the number of subjects with hepatitis c virus ribonucleic acid (HCV RNA) below a measurable laboratory limit, 12 weeks after completing therapy.
Time Frame: 12 weeks after completing treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure Cohort | Lung Disease Cohort
Number analyzed (Participants) | 10 | 5
Participants | 10 | 3
Statistical Analysis 1: Comparison: Heart Failure Cohort vs Lung Disease Cohort; Test type: Other; Proportion = 86.7, 95% CI 2-sided [59.5 to 98.3]

3. Secondary Outcome: Number of Subjects With Sustained Virologic Response (SVR) 4
Description: The secondary outcome of efficacy will be determined by the number of subjects with hepatitis c virus ribonucleic acid (HCV RNA) below a measurable laboratory limit, 4 weeks after completing treatment.
Time Frame: 4 weeks after completing treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure Cohort | Lung Disease Cohort
Number analyzed (Participants) | 10 | 5
Participants | 8 | 3

4. Other Pre Specified Outcome: Discontinuation for Adverse Events and Serious Adverse Events
Description: Assessment for discontinuation due to adverse events and serious adverse events, as addressed by adverse events and laboratory tests. Final study visit is 12 weeks after treatment.
Time Frame: 12 weeks after completing treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Failure Cohort | Lung Disease Cohort
Number analyzed (Participants) | 10 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 36 weeks
Arm/Group | Heart Failure Cohort | Lung Disease Cohort
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT02858180/Prot_SAP_000.pdf